CLINICAL TRIAL: NCT03403179
Title: A Pilot Study of Functional Remediation for Bipolar Disorder: Feasibility and Preliminary Efficacy
Brief Title: Functional Remediation for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sagar Parikh, Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00113668
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Bipolar Disorder
Keywords: Cognition; Cognitive Remediation; Mood Disorder; Functional Impairment; Psychosocial intervention
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders

STUDY DESIGN:
Intervention Model Description: This study is a single center, open-label, outpatient clinical trial with no randomization or blinding. The Barcelona Functional Remediation for Bipolar Disorder (FR) Program will be tested over a 21-week period using 30 participants split into two equal cohorts. The study will evaluate the feasibility and preliminary efficacy of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving Psychosocial Intervention (Experimental): Functional Remediation: The functional remediation program consists of 21 weekly sessions, each lasting 90 min. This intervention addresses neurocognitive issues such as attention, memory and executive functions, but it focuses even more on enhancing functioning in daily routine. The content of the intervention is based on ecological tasks to be performed in two settings, in the clinic as well as at home. Participants will be trained with exercises for memory, attention, problem solving and reasoning, multitasking and organization in order to improve their functional outcome. Most of the techniques are based on paper-and-pencil tasks and group activities.
  Interventions: Other: Functional Remediation

INTERVENTIONS:
Other: Functional Remediation — Functional Remediation: The functional remediation program consists of 21 weekly sessions, each lasting 90 min. This intervention addresses neurocognitive issues such as attention, memory and executive functions, but it focuses even more on enhancing functioning in daily routine. The content of the intervention is based on ecological tasks to be performed in two settings, in the clinic as well as at home. Participants will be trained with exercises for memory, attention, problem solving and reasoning, multitasking and organization in order to improve their functional outcome. Most of the techniques are based on paper-and-pencil tasks and group activities.

SUMMARY:
Bipolar Disorder is a major mood disorder with periodic mood episodes that may be very distressing, both to the individual and to others. When ill, the person is at particular risk for disruptions to social and occupational functioning, physical health, and even premature death. When not in an episode, individuals with BD may still be feeling well but have ongoing neurobiological processes, as well as the psychological sequelae from illness episodes, that can lead to subtle neurocognitive impairment that impedes overall functioning. This study is a test of an existing, published intervention that ameliorates deficits in functioning in euthymic bipolar individuals.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bipolar I or II disorder (BD), as determined by a structured diagnostic interview
* at least three months of clinical remission (euthymia or minimal symptoms), based on the phone screen assessing mood episodes in the prior three months
* score greater than 11 on a measure of everyday functioning (FAST; described in measures section) indicating at least mild impairment
* use of a standard bipolar mood-stabilizing medication at the same, adequate dose (according to CANMAT treatment guidelines) for at least 3 months prior to screening, with ability to continue that dose during the study.

Exclusion Criteria:

* history of neurological illness or injury (e.g., stroke, brain tumor)
* documented intellectual disability
* inability to provide written informed consent
* substance dependence within last 3 months or substance abuse in last 30 days
* inability to complete the six-month intervention
* received ECT in the past 12 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Feasibility | 30 weeks
  Feasibility will be determined by a composite of ability to recruit and deliver the treatment intervention to both cohorts of participants, with adequate delivery of the intervention as measured by completion of the manual's objectives.
Acceptability (Subject Satisfaction) | 30 weeks
  Acceptability of the intervention will be measured by use of the Satisfaction with Therapy and Therapist Scale.
Acceptability (Subject completion) | 30 weeks
  Measured by percentage of subjects who complete the intervention.

SECONDARY OUTCOMES:
Functional Impact | 30 weeks
  The Functioning Assessment Short Test (FAST) is an interviewer-administered scale for disability due to psychiatric illness, used both pre-and post-completion. The instrument has 24 items capturing 6 domains of functioning: (1) Autonomy (2) Occupational Functioning (3) Cognitive Functioning (4) Financial Issues (5) Relationships (6) Leisure Time. Scores above 11 identify at least mild functional impairment. Impact of the intervention on change in FAST score will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Parikh, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Depression Center, Ann Arbor, Michigan, United States